CLINICAL TRIAL: NCT03403998
Title: Effectiveness of Neck Motor Control Exercises in Patients With Temporomandibular Disorders: A Pilot Randomized Controlled Trial
Brief Title: Neck Exercises in Patients With Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00073078
Record Dates: First submitted 2018-01-03; First posted 2018-01-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Temporomandibular Disorders; Temporomandibular Joint Pain
Keywords: Pain; Temporomandibular Disorders; Therapeutic exercises; Musculoskeletal disorders; Randomized controlled trial; Imaging; Brain plasticity; Clinical outcomes; Chronic pain; Neck
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain; Musculoskeletal Diseases; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomization sequence will be computer-generated by a research assistant (RA) not involved in the study. To ensure concealment, the RA will distribute the results of the sequence to the therapist in consecutively numbered, opaque, and sealed envelopes. Participants will be unaware of the study hypothesis. Assessors (who will measure clinician-assessed tests and analyze imaging outcomes) and the statistician will be blinded to the hypothesis and group allocation, following established guidelines. Participants randomized to the treatment group will receive MCTF as described in the Intervention section. Participants randomized to the placebo group will receive placebo transcutaneous electrical nerve stimulation (TENS) as described in the Intervention section
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients (reporting one of the main outcome for this study - pain) will be unaware of the hypothesis of this study and performance biases will be avoided by telling them that both treatment options have similar effectiveness. Assessors (measuring clinician assessed tests) and Statistician will be blinded to hypothesis and group allocation following established guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises (Experimental): Neck flexors Training: Each patient will initially perform cranio-cervical flexion to sequentially reach 5 pressure targets in 2 mmHg increments from a baseline of 20 mmHg to the final level of 30 mmHg. For each target level, the contraction duration will be increased to 10 s, and the participant trained to perform 10 repetitions with brief rest periods between each contraction. Once one set of 10 repetitions of 10 s is achieved at one target level, the exercise will be progressed to train at the next target level up to the final target. Neck extensors training: Patients will perform cranio-cervical extension and upper cervical rotation in a prone on elbows position while maintaining the cervical spine in a neutral position, progressing to a 4-pt kneeling position.
  Interventions: Other: Exercises
- Placebo (Placebo Comparator): The placebo group will receive placebo TENS (switched-off TENS apparatus with no perceptible stimulation). Four electrodes, 50 x 35 mm, will be placed on the neck muscles. The participant will be informed that this therapy is called a "subthreshold current" and they might not be able to feel any sensation underneath the electrodes during the treatment. The placebo treatment will be for 30 min twice a week for 8 weeks, as for the intervention group.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Exercises — The treatment will consist of an 8-week progressive exercise program of neck flexors and extensors exercises supervised by a physical therapist for 30-45 min twice a week per 8 weeks as described in Arm/group descriptions.
  Arms: Exercises
Other: Placebo — The placebo treatment will be for 30-45 min twice a week for 8 weeks, as for the intervention group. ( see details in arm description)
  Arms: Placebo

SUMMARY:
Musculoskeletal (MSK) pain is a common reason to seek medical treatment. Temporomandibular disorders (TMDs) are MSK disorders that affect the masticatory muscles, the temporomandibular joint, and related structures in the neck and head. Current research showed that people with chronic TMDs have structural and functional brain changes that may contribute to chronic pain development and maintenance. Therapeutic exercise is a central component in treating chronic MSK conditions. New therapies, including exercise, appear to have potential in targeting cortical changes to improve clinical outcomes. However, mechanisms of action are not well understood, and evidence is limited to a few weak studies and specific populations. Evidence from our research group highlights neck exercise as potentially useful in treating TMDs. However, we do not yet know how the brains of women with TMD respond to specific exercise and whether these changes relate to decreased pain, improved function, and quality of life. Evidence linking brain plasticity, pain modulation, and exercise therapy is currently limited, and non-existent for people with TMDs. Objectives: In women with chronic TMD pain, we will:1) determine the impact of motor control training using visual feedback (MCTF) on clinical outcomes such as pain intensity and jaw disability, 2) assess the impact of MCTF on brain structure, using diffusion tensor imaging, 3) assess the impact of MCTF on brain networks, using resting state functional magnetic resonance imaging, and 4) determine the effectiveness of MCTF to restore normal muscular structure, performance and fatigability of neck cervical muscles, using electromyographic analysis. Methods: Women with chronic TMD pain will be randomized to either an intervention arm or a placebo control group. Women in the intervention arm will receive 8 weeks of progressive exercise MCTF of the cervical muscles, twice per week. Women in the placebo arm will receive innocuous transcutaneous electrical nerve stimulation (turn off). Our primary outcomes will be changes in 1) pain, measured with the Visual Analogue Scale, 2) brain structure and networks, measured by fractional anisotropy (brain structure) and the blood-oxygen-level dependent signal (brain networks). Outcomes will be measured at baseline, after 8 weeks of treatment, and 4 months after treatment ends. Results will directly inform and guide clinicians in prescribing more effective interventions for women with TMD

DETAILED DESCRIPTION:
To treat musculoskeletal disorders, looking at the brain is an unusual strategy but one with high potential for effectiveness. Exercise can potentially train the brain if we understand the links between exercise and productive changes in the brain. Given the high prevalence, impact, and burden of musculoskeletal disorders (MSKDs), therapies need to focus on the origin of the problem to be more effective and reduce economic costs. The latest evidence highlights the need for musculoskeletal rehabilitative therapy, including exercise, to look both at local structural and functional abnormalities of the MSK system and at alterations within the central nervous system. These central alterations have been shown to have a crucial role in the pathophysiology and clinical manifestations of MSKDs. People with chronic MSKDs show brain alterations such as decreased regional grey matter volume in brain areas such as the cingulate cortex, the insula, and the superior frontal and temporal gyrus. They also have impairments in pathways related to pain modulation. These brain alterations are visible in people with chronic MSKDs such as low back pain, osteoarthritis, headaches, and chronic temporomandibular disorders (TMDs).

Therapeutic exercise is a cornerstone for MSKD rehabilitation. Although its effects on pain are not fully understood, therapeutic exercise is widely applied in a variety of painful MSK conditions, including TMDs. Maladaptive changes in the motor cortex in MSKDs can improve after specific exercise training through motor control exercises and skilled cognitive practice, through strength and resistance training, and through novel motor training and visual feedback. However, all this evidence comes from preliminary studies with small sample sizes, before-and-after designs, and in specific clinical populations. Expanding this knowledge base to other clinical populations, with stronger study designs such as randomized controlled trials (RCTs), is important to accurately understand the effects of exercise therapy on brain plasticity and determine whether this approach is effective to manage MSKDs.

Our team is interested in managing TMDs through exercise therapy. From our previous studies on neck muscle impairment in people with TMDs and our recent update of a systematic review on therapeutic exercise to manage TMDs, we conclude that motor control exercise is a promising option to treat people with TMDs. However, the evidence is still limited and more high-quality investigations on the effectiveness of novel motor training in TMDs is needed.

OBJECTIVES

1. Determine the impact of motor control training using visual feedback (MCTF) on pain-disability related outcomes such as pain intensity, pain pressure thresholds and jaw disability. We will compare outcomes for people with TMDs who receive MCTF or a placebo treatment after 8 weeks of treatment, and 4 months after treatment ends.
2. Assess the impact of MCTF and explore its mechanisms of action on brain structure using DTI.
3. Assess the impact of MCTF on brain networks using rsfMRI.
4. Determine the effectiveness of MCTF in people with TMDs to restore normal muscular structure, performance and fatigability of the cervical muscles when compared with a placebo group.

THE PROPOSED TRIAL: MATERIALS AND METHODS Design: This study will be a randomized controlled trial (RCT). A randomization sequence will be computer-generated by a research assistant (RA) not involved in the study. To ensure concealment, the RA will distribute the results of the sequence to the therapist in consecutively numbered, opaque, and sealed envelopes. Participants will be unaware of the study hypothesis. Assessors (who will measure clinician-assessed tests and analyze imaging outcomes) and the statistician will be blinded to the hypothesis and group allocation, following established guidelines. Participants randomized to the treatment group will receive MCTF as described in the Intervention section. Participants randomized to the placebo group will receive placebo transcutaneous electrical nerve stimulation (TENS) as described in the Intervention section.

Participants: A convenience sample of people who attend the TMD/Orofacial Pain clinic (School of Dentistry, Faculty of Medicine & Dentistry, University of Alberta (UofA)) will be recruited.

Sample Size: This will be a pilot study. Based on data of previous study, using pain intensity as a main outcome and the ANOVA repeated measures within-between interaction (effect size d=0.27) using α=0.05 and β=0.95, a sample size of approximately 18 subjects per each group is required. Due to the possibility of a 10% of dropouts, we will recruit 20 subjects per group. Sample size calculation for the MRI variables was based on values of FA measurements of White Matter (WM) obtained from the WM adjacent to S1/M1 area obtained from Moayedi et al study on subjects with TMD. Based on a moderate difference between groups (effect size d=0.7) using α=0.05 and β=0.20, using an ANOVA analysis for 2 groups, a sample size of approximately 10 subjects per each group is required

PROCEDURES General Considerations: An experienced assessor will determine eligibility of participants and will evaluate them with the standardized forms from the new DC/TMD. REDcap, a password protected web platform (supported by the UofA) will be used to collect all outcomes.

Twenty subjects (10 subjects from the exercise group and 10 subjects from the placebo group) will be randomly allocated to undergo magnetic resonance imaging assessments of their brains at baseline, 2, and 6 months after randomization for both groups (treatment and control groups) if budget permits.

Primary Outcome Variables: The main outcome measures for this study are pain intensity (measured by the VAS) and Fractional Anisotropy (FA) and functional brain networks (evaluated by imaging).

All MRI will be performed in the Peter S. Allen MR Imaging Centre at the UofA by a certified MRI technologist.

Secondary Outcomes: will be discussed in the section of outcomes. The following will be considered secondary outcomes: The Neck Disability Index, Jaw function, Pressure pain threshold (PPT), cervical flexor muscle performance, Neck Extensor Endurance Test (NEET), the Neck Flexor Endurance test (NFET), Neck muscle structure, and Global Rating Scale (GRS)

INTERVENTION Early evidence from our research has shown that participants with TMDs present with abnormalities of the cervical flexor and extensor muscles. Exercises targeting these impairments reduce pain and level of dysfunction in people with cervical involvement. Thus, cervical motor control exercises are one of the most promising choices to treat people with TMDs. Treatment will consist of an 8-week progressive program of neck flexor and extensor exercises, performed for 30-45 min twice a week.

Neck flexor training: Exercise during the first stage will be an incremental craniocervical flexion movement in a relaxed, supine lying position. This exercise targets the deep flexors of the upper cervical region, the longus capitis and colli, rather than the superficial flexors, the sternocleidomastoid and anterior scalene muscles. Participants will be instructed to perform and hold progressively inner range positions of craniocervical flexion, using a pressure biofeedback connected to a screen. This will maximize feedback to the participants as described in Armijo-Olivo et al. Once the correct craniocervical flexion motion is achieved, participants will begin to hold progressively increasing ranges of craniocervical flexion. They will use feedback from the pressure unit placed behind their neck for 5 pressure targets (from 20 mmHg to 30 mmHg). Participants will be asked to hold each level for 10 s and perform 10 repetitions without compensatory movements, with brief rest periods between each contraction (~3-5 s). In the last 2 weeks of the exercise program, participants will perform higher-load exercise with head weight as the load. Numbers of repetitions and sets will be increased as permitted by the participant's response to the exercise. An endurance element will be incorporated by increasing the time the position is held, depending on the participant's progress.

Neck extensor training: Initially, participants will perform craniocervical extension and upper cervical rotation in a prone on elbows position while maintaining the cervical spine in a neutral position. They will progress to a 4-pt kneeling position. These exercises are designed to target the sub-occipital muscles. Attention will first be given to the spinal and scapular postures in the prone on elbows or 4-pt kneeling position. In the second phase of the exercise program, participants will perform higher-load exercise with head weight as the load, focusing on training the deep cervical extensors (the semispinalis cervicis/multifidus group). In this stage, they will initially perform up to 15 repetitions of neck extension while maintaining their head in a neutral position during 4-pt kneeling. Numbers of repetitions and sets will be increased as permitted by the participant's response to the exercise. An endurance element will be incorporated by increasing the time the position is held, depending on the participant's progress.

Participants will be asked to refrain from seeking any additional treatment during the study and will be asked to register their compliance with the exercise program in a daily diary using REDCap.

Placebo: The placebo group will receive placebo TENS (switched-off TENS apparatus with no perceptible stimulation). Four electrodes, 50 x 35 mm, will be placed on the neck muscles. The participant will be informed that this therapy is called a "subthreshold current" and they might not be able to feel any sensation underneath the electrodes during the treatment. The placebo treatment will be for 30 min twice a week for 8 weeks, as for the intervention group.

STATISTICAL ANALYSIS The analysis will follow the intention to treat principle. We will test for significant differences in VAS, PPT, TMDs and neck disabilities at baseline, after 8 weeks of treatment, and 4 months after treatment ends (6 months) between participants receiving MCTF and a placebo group. A two-way mixed ANOVA with repeated measures will be used for each outcome (Objective 1); We will test for significant changes in FA at baseline, after 8 weeks of treatment, and 4 months after treatment ends (6 months) between participants receiving MCTF and a placebo group, using a two-way mixed ANOVA with repeated measures. To determine the relationship between FA and the pain-disability and psychological outcomes, a multiple regression analysis will be conducted (Objective 2); We will determine if there are significant changes in rsfMRI networks after 8 weeks of treatment, and 4 months after treatment ends (6 months) between individuals receiving MCTF and a placebo group, using a two-way mixed ANOVA with repeated measures for each outcome. To determine the relationship between rsfMRI and the pain-disability and psychological outcomes, a multiple regression analysis will be conducted (Objective 3); We will determine if there are significant changes in CCFT, NEET, and NEFT, and cervical muscle structure at baseline, after 8 weeks of treatment, and 4 months after treatment ends (6 months) between individuals receiving MCTF and a placebo group, using a two-way mixed ANOVA with repeated measures for each outcome (Objective 4).

Psychological functioning variables (distress, depression, anxiety) will be covariates. The alpha level will be set at α = 0.05. A Bonferroni adjusted p-value will be applied to correct for potential multiple comparisons and a Bonferroni post hoc test will be used to determine the significant difference between pairwise comparisons. Effect sizes and minimal important difference of the outcomes (using the GRS as an anchor measure) will be used to determine the clinical significance of results.

ELIGIBILITY:
Inclusion Criteria:

1. females 18-60 years of age (TMDs are more prevalent in females);
2. diagnosed with muscle pain disorders as classified by the new Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) or mixed TMD;
3. have had pain in the masticatory muscle for at least 3 months;
4. have chronic masticatory muscle pain not attributable to recent acute trauma, previous infection, or active inflammation; and
5. have a moderate or severe baseline pain score of 30 mm or greater using a 100 mm VAS.

Exclusion Criteria:

1. metabolic, rheumatoid, or vascular diseases;
2. commonly comorbid functional chronic pain disorders (e.g., irritable bowel syndrome, fibromyalgia);
3. psychiatric disorders (e.g., depression, schizophrenia);
4. abnormal neurological examination;
5. contraindication for MRI scanning (e.g., metallic surgical implant);
6. self-report of substance abuse;
7. exercise therapy in the 6 months before entry into the study or current treatment for TMD;
8. previous experience with electrotherapy; or
9. pregnant or planning a pregnancy.

After confirming eligibility to participate in the study, all participants will be asked to sign an informed consent in accordance with the UofA´s policies on research using human participants.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity measured with a Visual Analogue Scale (VAS) | Change from baseline at 2 months ( change from baseline at 6 months )
  The VAS is a linear scale 10 cm in length, labeled with the two extremes boundaries of pain sensation: "no pain", at one end and "worst pain imaginable" at the other end. The validity and reliability of these methods for determining pain intensity, has been reported and confirmed in the literature
Fractional Anisotropy (FA) | Change from baseline at 2 months (change from baseline at 6 months (if budget allows))
  To analyze the DTI images, we will use a method similar to Moayedi et al. To analyze the rsfMRI images, we will use the pipeline outlined in Greicius et al.in addition to applying functional connectivity (graphical modelling) as previously used in our lab. Images will be imported into the software library (FSL v. 4.1.8) of the Oxford Centre for Functional MRI of the Brain (FMRIB). Preprocessing will include current and motion artifact correction using the FMRIB Diffusion Toolbox v. 2.0. The DTI images will be processed through 2 different pipelines for 1) voxel-wise analysis and 2) tractography. The preprocessed images will be fit with a diffusion tensor model using DTIFIT in the FDT. We then will calculate voxel-wise values of FA. The rsfMRI images will be analyzed using an ICA approach to isolate the DMN and the sensorimotor network and a functional connectivity approach using graphical modelling to assess the neural networks associated with TMD treatment.
functional brain networks | Change from baseline at 2 months (change from baseline at 6 months (if budget allows))
  To analyze the DTI images, we will use a method similar to Moayedi et al. To analyze the rsfMRI images, we will use the pipeline outlined in Greicius et al.in addition to applying functional connectivity (graphical modelling) as previously used in our lab. Images will be imported into the software library (FSL v. 4.1.8) of the Oxford Centre for Functional MRI of the Brain (FMRIB). Preprocessing will include current and motion artifact correction using the FMRIB Diffusion Toolbox v. 2.0. The DTI images will be processed through 2 different pipelines for 1) voxel-wise analysis and 2) tractography. The preprocessed images will be fit with a diffusion tensor model using DTIFIT in the FDT. We then will calculate voxel-wise values of FA. The rsfMRI images will be analyzed using an ICA approach to isolate the DMN and the sensorimotor network and a functional connectivity approach using graphical modelling to assess the neural networks associated with TMD treatment.

SECONDARY OUTCOMES:
Jaw function | Change from baseline at 2 months ( change from baseline at 6 months )
  Will be measured using a self-reported questionnaire called "Limitations of Daily Functions in TMD Questionnaire" (LDF-TMDQ/JFS, available upon request).The internal consistency of this questionnaire is high and there is good convergent validity with the dental version of the McGill Pain Questionnaire.The total score of the questionnaire summing the patient's answers will be used for statistical purposes.
Neck Flexor Endurance Test | Change from baseline at 2 months ( change from baseline at 6 months )
  The subjects will be asked to perform a maximal isometric cervical extension contraction (MVC) (for 5 seconds). Once the tester has ensured that the subject has learned the procedure, each subject will be asked to perform the maximal voluntary isometric contraction (MVC). Each subject will perform 2 repetitions of this movement allowing 5 minutes between each trial to avoid fatigue. The average force value of the 2 contractions will be used as the reference MVC. This will allow submaximal target contractions (25% MVC) to be set on the visual feedback display related to this value. After performing the MVC, and when the tester has ensured that the subject had learned the procedure for doing submaximal contractions with the help of the visual biofeedback, each subject will be asked to perform 2 submaximal cervical flexion contractions at 25% MVC, keeping the chin retracted, and maintain these contractions if possible using a visual display for feedback of the force output.
Neck Extensor Endurance Test: | Change from baseline at 2 months ( change from baseline at 6 months )
  Subjects will be asked to perform a maximal isometric cervical flexion contraction (MVC) (for 5 seconds). Each subject will perform 2 repetitions of this movement allowing 5 minutes between each trial to avoid fatigue. The average force value of the 2 contractions will be used as the reference MVC. This will allow submaximal target contractions (25% MVC) to be set on the visual feedback display related to this value. After performing the MVC, and when the tester has ensured that the subject had learned the procedure for doing submaximal contractions with the help of the visual biofeedback, each subject will be asked to perform 2 submaximal cervical flexion contractions at 25% MVC, keeping the chin retracted, and maintain these contractions as long as possible using a visual display for feedback of the force output.
Craniocervical Flexion Test (CCFT) | Change from baseline at 2 months ( change from baseline at 6 months )
  CCFT is performed using a pressure biofeedback device located in the neck region, and a visual aid positioned in front of the subject, with the subject lying supine, keeping the legs flexed. Each subject will be attempted to reach 5 different levels. The device will have a graduation with marks corresponding to increments of 2mmhg, ranging from 20mmhg to 30mmhg. The level of effort required in the test will be progressive, and observed according to what the subject can perform. To move to the next level, the subject must be able to complete ten 10-second repetitions on each possible level. When the subject starts to use the superficial musculature or to do some compensation of the movement, it will be time to finish the test. The cumulative performance Index (CPI) will be calculated. A perfect CPI of 300 will be obtained if the participant could progress through all levels without showing signs of compensations and/or fatigue.
Global Rating Scale (GRS) | Change from baseline at 2 months ( change from baseline at 6 months )
  All Subjects will be asked to rate the change they have experienced in jaw pain and jaw function before and after the treatment using a global rating scale (GRS). This scale can be used by subjects to rate the magnitude of change they have experienced, in this case, after the exercise therapy at two and at six months. Subjects will identify the degree of change by responding on a 15-point Likert scale, with -7 = a very great deal worse, 0 = about the same, and +7 = a very great deal better.
The Neck Disability Index | Change from baseline at 2 months ( change from baseline at 6 months )
  Is a 10-item questionnaire that measures how much neck pain affects activities of daily living such as personal care, lifting, reading, headaches, concentration, work, driving, and sleeping. The NDI is a validated, reliable and responsive relatively short questionnaire that can be easily administered. For the purpose of this study, the total score of the questionnaire summing the patient's answers was used for statistical purpose.
Psychological functioning: distress | Change from baseline at 2 months ( change from baseline at 6 months )
  will be measured by the questionnaire recommended by the DC/TMD: patient health questionnaire-4 (PHQ-4) for distress
Pressure Pain Threshold (PPT) | Change from baseline at 2 months ( change from baseline at 6 months )
  Pressure pain sensitivity (PPS) is the most commonly used method for quantitative analysis of local muscle pain and tenderness in pain research. PPS will be evaluated via pressure pain threshold (PPT), or the minimum pressure that induces pain or discomfort. This will be done in the masticatory muscles and neck muscles using a calibrated mechanical algometer (Wagner Instruments, Greenwich, CT 06836-1217) following the protocol described in Silveira et al. PPT measurements have been shown to have good or excellent inter-rater and intra-rater reliability (0.74 to 0.99).
Muscle structure | Change from baseline at 2 months ( change from baseline at 6 months )
  Muscle structure will be measured through MRI assesment
Psychological functioning: depression | Change from baseline at 2 months ( change from baseline at 6 months )
  depression will be measured by the patient health questionnaire-9 (PHQ-9) for depression,
Psychological functioning: anxiety | Change from baseline at 2 months ( change from baseline at 6 months )
  Anxiety will be measured by the general anxiety disorder-7 (GAD-7) instrument.
therapeutic alliance | at 2 months
  The therapeutic alliance between the therapist and the patient will be measured at 1 month and at the end of the treatment by using the working alliance sub-scale of the Pain Rehabilitation Expectations Scale (PRES). The PRES is a self-reported clinical intervention-specific assessment tool developed to measure proxy efficacy, motivation/ expectations, and working alliance for rehabilitation interventions in LBP patients
level of expectations | baseline
  Patients will be asked to rate their expectations of pain relief at baseline using the Credibility and Expectancy Questionnaire (CEQ). The CEQ tool has been widely used in clinical trials in diverse areas such as psychology (66,67) pharmacology (68) physiotherapy (69), and cognitive-behavioral therapy (70) to determine level of expectations. The CEQ comprises 6- items (2 sets) and two factors (i.e. credibility and expectancy). Items 1 to 3 measure credibility, while items 4 to 6 appraise expectancy. Subjects are asked to rate items on a scale of 1 to 9, with anchors provided for 1 ("not at all), 5 ("somewhat"), and 9 ("very"). Thus, for the expectancy variable a minimum score of 3 points and a maximum of 27 points can be obtained. The CEQ is considered to be a valid and reliable (71) tool to measure the expectancy construct.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Armijo-Olivo, PhD, Principal Investigator — University of Alberta
Locations (1):
- Corbett Hall-Sports Laboratory, Edmonton, Alberta, Canada